CLINICAL TRIAL: NCT04862728
Title: Role of Various Nutritional Interventions in Management of Critically Ill Child
Brief Title: Role of Nutritional Intervention in Critically Ill Child
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hanan Saad Ahmed Hamdallah, principle investigator, Assiut University
Other Study IDs: malnutrition in critically ill
Record Dates: First submitted 2021-04-17; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Nutrition Disorder, Child
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: - Strong kids screening tool - Stamp screening tool - PYMS screening tool — Screening Tool for the Assessment of Malnutrition in Pediatrics (STAMP) evaluates patient's clinical diagnosis, nutritional intake during hospitalization and anthropometric measurements, developing a care plan based on the child's overall malnutrition risk (low, medium or high).Screening Tool for Impaired Nutritional Status and Growth (STRONG kids). It consists of four items: subjective clinical assessment, high-risk diseases, nutritional intake and losses, weight loss or poor weight gain. Patients classified at high nutritional risk have a longer hospitalization and a negative standard deviation score (SDS) for weight-for-height (WFH), which indicated a state of acute malnutrition.The Pediatric Yorkhill Malnutrition Score (PYMS) is adopted among medical and surgical patients between 1 and 16 years of age. The PYMS assesses four items: BMI, history of recent weight loss,
  Other Names: early versus late enteral nutrition on the outcome and predict complication.

SUMMARY:
* Assess the nutritional status of critically ill children using different nutritional assessment tools in management.
* Assess accuracy and validity of screening tools in diagnosis of malnutrition by the following:

  * Strong kids
  * Stamp
  * PYMS
* Assess the effect of early versus late enteral nutrition on the outcome and predict the complication associated with enteral feeding.

DETAILED DESCRIPTION:
Malnutrition affects millions of children throughout the World. According to ESPEN nutritional risk screening tools have been designed to detect protein and energy under nutrition and predict if under nutrition may develop or worsen. The Screening was validated Tool for Assessment of Malnutrition in Pediatrics (STAMP) that evaluates patient's clinical diagnosis, nutritional intake during hospitalization and anthropometric measurements, developing a care plan based on the child's overall malnutrition risk. The Screening Tool for Impaired Nutritional Status and Growth (STRONG kids) consists of four items: clinical assessment, high-risk diseases, nutritional intake and losses, weight loss or poor weight gain.

The Pediatric Yorkhill Malnutrition Score (PYMS) is adopted among patients between 1 and 16 years of age assesses four items: BMI, history of recent weight loss, changes in nutritional intake and the expected effect of current medical condition on patient's nutritional status.

Indirect calorimetry, calculated from analysis of the inspired and expired gases, is the best method for evaluating individual energy expenditure.

Protein requirements are highe. The catabolic effects of illness lead to negative nitrogen balance. Randomized protein-supplemented enteral diet achieved 3.1g/kg/day protein and positive nitrogen balance by PICU day 5.

Enteral nutrition is more physiological, simpler, can be started more quickly and cheaper, it does not require special preparation, and it can be started and modified at any time.

Par enteral nutrition has reserved for those patients with intestinal obstruction or severe gastrointestinal damage, ischemia, inflammation, hemorrhage, peritonitis and paralytic ileus.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill children aged 1-5 years admitted to PICU.

Exclusion Criteria:

* Infants before the age of one year and children after the age of five years.
* Any child with chronic illness.
* Patients with multiorgans failure.
* Children with congenital anomalies.
* Children on renal dialysis.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study population will be taken from pediatric intensive care unit (PICU) at Assiut university Children Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Identifying high risk group of malnutrition among patient in PICU by nutritional assesement by Screening Tool for the Assessment of Malnutrition in Pediatrics. | baseline
  Screening Tool for the Assessment of Malnutrition in Pediatrics evaluates patient's clinical diagnosis nutritional intake during hospitalization and anthropometric measurements malnutrition risk. the measured value of the child's height and weight will recorded and compared to reference values by age. and gender
Identifying high risk group of malnutrition among patient in PICU by nutritional assesement by Screening Tool for Impaired Nutritional Status and Growth in kids. | baseline
  Screening Tool for Impaired Nutritional Status and Growth (STRONG kids) consists of subjective clinical assessment high risk diseases nutritional intake and losses. weight, poor weight gain Patients classified at high nutritional risk have a longer hospitalization and a negative standard deviation score for weight for height which indicated a state of acute malnutrition,this tool appeared rapid and easy to use, additionally it may predict long of hospital stay and identifies a need for nutritional interventions during the hospitalization.
Identifying high risk group of malnutrition among patient in PICU by nutritional assesement by The Pediatric Yorkhill Malnutrition Score. | baseline
  The Pediatric Yorkhill Malnutrition Score (PYMS) is adopted among patients between 1 and 16 years of age. It assesses BMI history of recent weight loss changes in nutritional intake and the expected effect of current medical condition on patient's nutritional status

SECONDARY OUTCOMES:
the importance of early versus late enteral nutrition for patient in PICU. | baseline
  We will conduct this study to compare early (6-24 h) with late (after 24 h) initiation of enteral feeding in PICU. Enteral nutrition is more physiological,early enteral nutrition has a trophic effect on the intestinal mucosa, and stimulates the intestinal immune system, decreasing bacterial overgrowth and translocation; it therefore reduces the incidence of sepsis and multiorgan failure. Furthermore,early enteral nutrition is associated with fewer hepatic and metabolic complications than late and parentral nutrition.

CONTACTS AND LOCATIONS:
Overall Officials: zenab Mohie EL Deen, professor, Study Chair — professor at pediatric departement, faculty of medecine, assiut university; Osama Al Asheer, professor, Study Director — professor at pediatric departement, faculty of medecine, assiut university; Amira Shalaby, lecturer, Study Director — lecturer at pediatric departement, fsculty of medicine, assiut university

REFERENCES:
- [Result] Hulst JM, Zwart H, Hop WC, Joosten KF. Dutch national survey to test the STRONGkids nutritional risk screening tool in hospitalized children. Clin Nutr. 2010 Feb;29(1):106-11. doi: 10.1016/j.clnu.2009.07.006. Epub 2009 Aug 13. PMID 19682776
- [Result] Gerasimidis K, Keane O, Macleod I, Flynn DM, Wright CM. A four-stage evaluation of the Paediatric Yorkhill Malnutrition Score in a tertiary paediatric hospital and a district general hospital. Br J Nutr. 2010 Sep;104(5):751-6. doi: 10.1017/S0007114510001121. Epub 2010 Apr 19. PMID 20398432
- [Result] McCarthy H, Dixon M, Crabtree I, Eaton-Evans MJ, McNulty H. The development and evaluation of the Screening Tool for the Assessment of Malnutrition in Paediatrics (STAMP(c)) for use by healthcare staff. J Hum Nutr Diet. 2012 Aug;25(4):311-8. doi: 10.1111/j.1365-277X.2012.01234.x. Epub 2012 May 9. PMID 22568534
- [Result] Joosten KF, Hulst JM. Nutritional screening tools for hospitalized children: methodological considerations. Clin Nutr. 2014 Feb;33(1):1-5. doi: 10.1016/j.clnu.2013.08.002. Epub 2013 Aug 31. PMID 24050847
- [Result] Skillman HE, Wischmeyer PE. Nutrition therapy in critically ill infants and children. JPEN J Parenter Enteral Nutr. 2008 Sep-Oct;32(5):520-34. doi: 10.1177/0148607108322398. PMID 18753390